CLINICAL TRIAL: NCT01408693
Title: Minimal Invasive Anterior Approach Versus Trans-gluteal Approach for Hemi-arthroplasty in Femoral Neck Fractures - A Prospective Randomized Trial
Brief Title: Minimal Invasive Anterior Approach Versus Trans-gluteal Approach for Hemi-arthroplasty in Femoral Neck Fractures
Acronym: MIS-CLAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHBS-TRAUMA-68/11
Record Dates: First submitted 2011-06-10; First posted 2011-08-03 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Femoral Neck Fracture
Keywords: hip fracture; hemiarthroplasty; endoprosthesis; elderly; minimally invasive surgery; anterior approach; geriatric patients
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anterior minimal invasive approach, AMIS (Active Comparator): AMIS in 95 randomized patients.
  Interventions: Procedure: Anterior minimal invasive approach, AMIS
- Trans-gluteal approach, CLAS (Active Comparator): CLAS in 95 randomized patients.
  Interventions: Procedure: Trans-gluteal approach, CLAS

INTERVENTIONS:
Procedure: Trans-gluteal approach, CLAS — Classic lateral, trans-gluteal approach. Device: Cemented unipolar hip hemiarthroplasty for the treatment of femoral neck fractures
  Other Names: Mecacta, Mathys, Switzerland
  Arms: Trans-gluteal approach, CLAS
Procedure: Anterior minimal invasive approach, AMIS — Minimal invasive Hueter anterior approach. Device: Cemented unipolar hip hemiarthroplasty for the treatment of femoral neck fractures
  Other Names: Medacta, Mathys, Switzerland
  Arms: Anterior minimal invasive approach, AMIS

SUMMARY:
The aim of the study is to test the hypothesis that patients older than 60 years with a femoral neck fracture eligible for hemi-arthroplasty (HA) operated by an anterior minimal-invasive approach as compared to a standard lateral Hardinge approach show better functional recovery postoperatively as measured by the "Timed up and go"-test (TUG).

DETAILED DESCRIPTION:
HA via various well established approaches is the typical treatment for displaced femoral neck fractures in elderly patients. In the last decade, so called minimal-invasive surgery (MIS) for the implantation of total hip arthroplasty (THA) has become popular and studies have demonstrated that MIS is as safe as conventional approaches. Our hypothesis is that femoral neck fracture patients may especially benefit from MIS. To date, no published data exist comparing a Hueter minimal-invasive anterior (AMIS) with a conventional trans-gluteal Hardinge approach (CLAS) for HA.

Geriatric patients presenting at the University hospital Basel (UHBS) with a femoral neck fracture eligible for HA are randomly assigned to the minimal-invasive or conventional group. In both groups HA will be performed using the same implants. Postoperatively patients will be followed-up continuously until discharge from our hospital (with 7 days as expected average duration of postoperative hospital stay) with a first functional status assessment on day 5. Further follow-up is planned at week 3 and 6, 3 months and one year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age of 60 years or more, ambulatory with/without walking aids before trauma
* Femoral neck fracture eligible for hemi-arthroplasty in accordance with the algorithm for femoral neck fracture patients used at the University hospital Basel
* Informed consent

Exclusion Criteria:

* Refusal of consent by the patient or legal representatives to participate in the study
* More than one fracture
* Suspicion of a pathological fracture in the context of known or unknown malignancy
* Previous surgery of the proximal femur on the same side
* Follow-up not possible (Tourist etc.)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2011-08; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Timed up and go test (TUG) | 3 weeks postoperatively +/- 3 days
  TUG: Time in seconds a person needs to stand up from a chair, walk a distance of 3 meters, turn around a flag, come back and sit down again (with or without walking aids).

SECONDARY OUTCOMES:
Functional Independence measure (FIM) | preoperative (retrospective assessment), day 5 postoperatively, 3 and 6 weeks postoperatively, 3 months and 1 year postoperatively (apart from measurement on day 5 postoperative each +/- 3 days )
  FIM is a widely used method of assessing quality of daily life and the amount of assistance required for a person with a disability to perform basic activities safely and effectively. It includes 18 items focusing on a minimum set of skills related to self-care, sphincter control, transfers, locomotion, communication, and social cognition. Possible scores range from 18 to 126.
Postoperative complications | duration from surgery until 1 year postoperatively
  Postoperative complications (proximal femoral fracture, nerve palsy, postoperative surgical site infection, aseptic loosening, peri-prosthetic fracture, re-operation, non-surgical complications etc.) as a secondary outcome variable will be continuously recorded using the Clavien-Dindo classification of surgical complications
Peri-operative delirium | duration from admission to day 3, an expected average period of 3-5 days
  To assess delirium, patients will be screened 3 times a day by the responsible nurse using a modified Delirium Observation Screening scale (DOS). DOS is a 13-item scale for early recognition of delirium. If DOS results in equal or more than 3 points, the Confusion Assessment Method (CAM) will be additionally applied. The CAM instrument consists of 4 respectively 5 operationalized criteria from the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).
One year mortality | one year
Length of hospitalization | duration of the hospital stay, an expected average of 10 days
Subgroup effect of patients with normal Mental-state Questionnaire (MSQ) versus patients with abnormal (MSQ) | one year
  Corresponding to the results of the mental state questionnaire at the admission patients are evaluated able to judge or not able to judge. An analysis of subgroup-effect for the other outcome variables will be done.
Peri-operative factors | Peri-operative period, i.e. time between admission until day 5 postoperative, expected average period of 5-8 days
  Blood loss (estimated by anesthesiologist and surgeon) and blood transfusion (amount) Duration of surgery (skin-incision - skin closure)
Timed up and go test (TUG) | day 5, 6 weeks, 3 month and 1 year postoperatively (each +/- 3 days)
  see primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Jakob, Professor, Principal Investigator — Department of Traumatology, University hospital Basel
Locations (1):
- Department of Traumatology, University Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Keith RA, Granger CV, Hamilton BB, Sherwin FS. The functional independence measure: a new tool for rehabilitation. Adv Clin Rehabil. 1987;1:6-18. No abstract available. PMID 3503663
- [Background] Schuurmans MJ, Shortridge-Baggett LM, Duursma SA. The Delirium Observation Screening Scale: a screening instrument for delirium. Res Theory Nurs Pract. 2003 Spring;17(1):31-50. doi: 10.1891/rtnp.17.1.31.53169. PMID 12751884
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Matta JM, Shahrdar C, Ferguson T. Single-incision anterior approach for total hip arthroplasty on an orthopaedic table. Clin Orthop Relat Res. 2005 Dec;441:115-24. doi: 10.1097/01.blo.0000194309.70518.cb. PMID 16330993
- [Background] Rachbauer F, Kain MS, Leunig M. The history of the anterior approach to the hip. Orthop Clin North Am. 2009 Jul;40(3):311-20. doi: 10.1016/j.ocl.2009.02.007. PMID 19576398
- [Background] Smith TO, Blake V, Hing CB. Minimally invasive versus conventional exposure for total hip arthroplasty: a systematic review and meta-analysis of clinical and radiological outcomes. Int Orthop. 2011 Feb;35(2):173-84. doi: 10.1007/s00264-010-1075-8. Epub 2010 Jun 18. PMID 20559827
- [Derived] Saxer F, Studer P, Jakob M, Suhm N, Rosenthal R, Dell-Kuster S, Vach W, Bless N. Minimally invasive anterior muscle-sparing versus a transgluteal approach for hemiarthroplasty in femoral neck fractures-a prospective randomised controlled trial including 190 elderly patients. BMC Geriatr. 2018 Sep 21;18(1):222. doi: 10.1186/s12877-018-0898-9. PMID 30241509